CLINICAL TRIAL: NCT06267456
Title: The Reliability of Upper Extremity Rotation Test in Overhead Athletes and Its Relationship With Selected Upper Extremity Performance Tests
Brief Title: The Reliability of ULRT in Overhead Athletes and Its Relationship With Selected UEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Research Assisstant, Sakarya Applied Sciences University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HÜ- FTR- BD- 01
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Upper Limb Asymmetry
Keywords: Physical performance test; shoulder; assessment

STUDY DESIGN:
Intervention Model Description: handball, volleyball and basketball players 18-30 years Someone who has been participating in sports for at least three years and trains at least three times a week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- handball players (Other): Handball players aged between 18 and 35 who have been playing for a minimum of 3 years.
  Interventions: Diagnostic Test: Upper Limb Rotation Test; Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Upper Quarter Y Balance Test
- volleyball players (Other): volleyball players aged between 18 and 35 who have been playing for a minimum of 3 years.
  Interventions: Diagnostic Test: Upper Limb Rotation Test; Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Upper Quarter Y Balance Test
- basketball players (Other): Basketball aged between 18 and 35 who have been playing for a minimum of 3 years.
  Interventions: Diagnostic Test: Upper Limb Rotation Test; Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Upper Quarter Y Balance Test

INTERVENTIONS:
Diagnostic Test: Upper Limb Rotation Test — The athlete is positioned with the shoulder, elbow lateral epicondyle, greater trochanter, and ankle lateral malleolus in contact with the wall. In the push-up position, the elbows are started at shoulder height with a 90° bend, and the feet are placed in a shoulder-width apart position. Athletes are instructed to perform a rotation of the shoulder and trunk by touching a vertically placed band on the wall for 15 seconds in the position of 90° abduction and 90° external rotation of the shoulder. The tested side is the upper extremity where the closed kinetic chain position is maintained.
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — Athletes were placed in a push-up position with a distance of 91.44 centimeters (cm) (3 feet) between their hands for the test position. Subsequently, they were instructed to touch one hand to the other as quickly as possible. The total number of touches within a 15-second period was recorded. Modified push-up position was used for women, and regular push-up position for men during this time. Prior to the test, a familiarization trial consisting of 5 repetitions was performed. The test was then repeated 3 times, and the average of these repetitions was recorded as the score. Individuals were given a 45-second rest period between repetitions. The normalized score, representing the touch count per individual's height, was calculated. The power score was obtained by multiplying the touch count by 68% of the individual's body weight in kilograms.
Diagnostic Test: Upper Quarter Y Balance Test — The Upper Extremity Y Balance Test was created using three rulers placed on the ground in the medial, inferolateral, and superolateral directions. The rulers in the superolateral and inferolateral directions were positioned at a 90° angle to each other, while the ruler in the medial direction was placed at a 135° angle with respect to these two directions. In this test, both arms started in a push-up position with shoulder-width apart. The athlete was then instructed to touch, using their non-dominant hand, the maximum reachable point in the medial, inferolateral, and superolateral directions.

SUMMARY:
Upper Extremity Rotation Test is a new test the evaluates 90-90 position, which is one of the requirements for overhead throwing. The aim of the study was to evaluate the reliability of the Upper Extremity Rotation Test in overhead athletes and the relationship between the Closed Chain Upper Extremity Stability Test and the Upper Quarter Y Balance Test.

DETAILED DESCRIPTION:
Upper Extremity Rotation Test is a new test the evaluates 90-90 position, which is one of the requirements for overhead throwing. The aim of the study was to evaluate the reliability of the Upper Extremity Rotation Test in overhead athletes and the relationship between the Closed Kinetic Chain Upper Extremity Stability Test and the Upper Quarter Y Balance Test. Upper Extremity Rotation Test was found to be reliable in overhead athletes. Upper Extremity Rotation Test showed high reliability in overhead atheletes. There was no correlation between the Upper Exremity Rotation Test and the Upper Quarter Y Balance Test. A moderate corelation was found between the Upper Extremity Rotation Test and Closed Kinetic Chain Upper Extremity Stability Test.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Continuing sports for at least three years for each group (volleyball, handball, baskeball)
* Athletes training at least three days per week.

Exclusion Criteria:

* Individuals experiencing difficulty understanding what the physiotherapist says.
* Having a history of orthopedic surgery within the last year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
The reliability of Upper Extremity Rotation Test | January 2022
  The reliability of the Upper Extremity Rotation Test was evaluated.

SECONDARY OUTCOMES:
The Relationship Assessment of the Upper Extremity Rotation Test | February 2022
  The relationship between the Upper Extremity Rotation Test and the Closed Kinetic Chain Upper Extremity Stability Test and Upper Quarter Y Balance Test was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül Dıngırdan, Master's, Principal Investigator — Sakarya Applied Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Birgül Dıngırdan, Kocaeli, İzmit
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No